CLINICAL TRIAL: NCT03958565
Title: Response of Bony Metastasis to Tyrosine Kinase Inhibitors in Non-Small Cell Lung Cancers With Actionable Driver Mutations
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Cancer League of Colorado (Other)
Responsible Party: Sponsor
Other Study IDs: 19-0392.cc; NCI-2019-03377 (Other: CTRP)
Record Dates: First submitted 2019-05-14; First posted 2019-05-22 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Tyrosine Kinase Inhibitors; Zoledronic Acid; Denosumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Actionable driver oncogene: One group will have an actionable driver oncogene and initiate treatment in any line with a TKI as standard of care and concurrent to participation to this study; expected to have an objective response rate in ≥40% who have not previously seen anti-bone resorptive therapy.
  Interventions: Biological: Tyrosine Kinase Inhibitor
- No Actionable Mutations: The other group will not have actionable mutations and initiate treatment with chemotherapy/immunotherapy along with new onset therapy with IV zoledronic acid 4mg Q4 weeks or subcutaneous denosumab 120 mg Q12 weeks for bone disease, which is standard of care and would be concurrent to participation in this study.
  Interventions: Drug: Zoledronic Acid 4 MG/100 ML Intravenous Solution [ZOMETA]; Drug: Denosumab 120 MG/1.7 ML Subcutaneous Solution [XGEVA]

INTERVENTIONS:
Biological: Tyrosine Kinase Inhibitor — Targeted therapy given as standard of care.
  Groups: Actionable driver oncogene
Drug: Zoledronic Acid 4 MG/100 ML Intravenous Solution [ZOMETA] — Given Q4 weeks as standard of care
  Groups: No Actionable Mutations
Drug: Denosumab 120 MG/1.7 ML Subcutaneous Solution [XGEVA] — Given Q12 weeks for bone disease as standard of care
  Groups: No Actionable Mutations

SUMMARY:
The purpose of this study is to assess percentage reduction in the of urine NTX and serum CTX , in patients with NSCLC and bone metastases 1) with actionable driver oncogene on standard of care (SOC) TKI at 3 months post treatment and 2) without actionable mutations on standard of care therapy (chemotherapy/immunotherapy) treated with zoledronic acid or denosumab at the same time period.

DETAILED DESCRIPTION:
This is an observational study involving two arms of NSCLC with metastatic bony disease at the time of enrollment in the study. One group will have an actionable driver oncogene and initiate treatment in any line with a TKI as standard of care and concurrent to participation to this study; expected to have an objective response rate in ≥40% who have not previously seen anti-bone resorptive therapy. The other group will not have actionable mutations and initiate treatment with chemotherapy/immunotherapy along with new onset therapy with IV zoledronic acid 4mg Q4 weeks or subcutaneous denosumab 120 mg Q12 weeks for bone disease, which is standard of care and would be concurrent to participation in this study.

Baseline and on-treatment imaging and serum total alkaline phosphatase will be performed per SOC.

Additional non-SOC bone turnover markers including , urine N-telopeptide (NTX) and serum C-terminal telopeptide (CTX), will be checked at baseline and then at 1, 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form
2. Stated willingness to comply with all study procedures and be available for the duration of the study
3. Be a male or female aged 18-100 years
4. Pathologically confirmed non-small cell lung cancer
5. Molecular testing through a CLIA-validated NGS assay. This can be done using either tissue based samples or blood-based samples (ctDNA)
6. ECOG PS 0-2
7. Decision to be on a particular standard of care TKI or chemotherapy +/- immunotherapy (clinical decision that would occur prior to study enrollment)
8. Patients who will be treated with an osteoclast inhibitor must receive dental clearance prior to starting treatment
9. Bone metastases must be detected through radiographic imaging prior to enrollment on this study.

Exclusion Criteria:

1. Actionable driver mutation NSCLC patient who has been on anti-bone resorptive therapy

   a. Excluded anti-bone resorptive therapy includes: zolendronic acid, pamidronate, alendronate, denosumab or any medication that acts as an osteoclast inhibitor
2. Have any condition or illness that, in the opinion of the investigator, would compromise participant safety or interfere with evaluation while on standard of care treatments for the NSCLC.
3. Patients with actionable driver mutation who received TKI in past or currently on TKI prior to screening
4. Bone metastases that have received prior radiotherapy unless unequivocal progression has occurred since radiation therapy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: About 30-40% of patients w/ lung cancer develop bone metastases during their disease; the median survival time of patients w/ this secondary lesion is 7 months. In a retrospective study of 259 non-small cell lung cancer (NSCLC) patients, the most common site of skeletal metastases was the spine in 50% of patients, followed by the ribs (27.1%), ilium (10%), sacrum (7.1%), femur (5.7%) &humerus, scapula & sternum (2.9%). At our institution, it is standard practice not to use anti-bone resorptive therapy in driver mutation-addicted NSCLC w/ bony metastasis, while anti-bone resorptive therapies are commonly used in NSCLC w/ bony metastases w/o any actionable driver mutation. This study relates to exploring the potential differential need for anti-resorptive bone medications (bisphosphonates or RANK-L inhibitors) in patients w/ advanced non-small cell lung cancer & bone metastases w/ & w/o actionable driver mutations.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-28 (Actual); Primary Completion 2028-03-05 (Estimated); Study Completion 2028-04-28 (Estimated)

PRIMARY OUTCOMES:
Percentage reduction of urine NTX and serum CTX | 3 months post-treatment
  The percentage reduction in the bone turnover markers including urine N-telopeptide (NTX) and serum C-terminal telopeptide (CTX) from baseline at 3 months from starting TKI (oncogene arm) or anti-resorptive therapy as part of standard systemic therapy (non-oncogene arm).

SECONDARY OUTCOMES:
Skeletal-related events (SREs) | 1, 3, 6, and 12 months post-treatment
  Skeletal-related events (SREs) defined as the adverse events associated with bone metastases. SREs would include pathologic fractures, the requirement for surgery or radiotherapy, spinal cord compression.
Progression Free Survival (PFS) | at 1 year
  Progression Free Survival (PFS) would be defined as progression of disease or death from any cause from time of randomization until the end of study.
Objective Response Rate (ORR) | at 1 year
  Objective Response Rate (ORR) defined as proportion of patients with reduction in bony metastases as evaluated by using both the MD Anderson (MDA) criteria for patients who receive CT or bone scans and Positron Emission Tomography Response Criteria in Solid Tumors (PERCIST) for patients who undergo FDG PET/CT. These criteria allow for categorization of disease response from complete response to progressive disease.
Percentage reduction in the bone turnover markers including urine N-telopeptide (NTX) and serum C-terminal telopeptide (CTX) | From Baseline at 1, 6, and 12 months post-treatment
  Percentage reduction in the bone turnover markers including urine N-telopeptide (NTX) and serum C-terminal telopeptide (CTX) from baseline at 1, 6 and 12 months.
Percentage normalization of blood total alkaline phosphatase | From baseline at 1, 3, 6, and 12 months
  Percentage normalization of blood total alkaline phosphatase from baseline at 1, 3, 6, and 12 months. Normal level of blood total alkaline phosphatase would be defined as equal or less than 147 IU/L.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Schenk, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Hospital, Aurora, Colorado
  - Lone Tree Medical Center, Lone Tree, Colorado

IPD SHARING:
Plan to Share IPD: Yes
Clinical data (including AEs, concomitant medications, and expected adverse reactions data) and clinical laboratory data will be entered into REDCap; the data system includes password protection and internal quality checks, such as automatic range checks, to identify data that appear inconsistent, incomplete, or inaccurate. Clinical data will be entered directly from the source documents.Data will be tracked using REDCap. Data collected for this study will be analyzed and stored at the University of Colorado Cancer Center.
  When the study is completed, access to study data will be provided through the UCCC Oncology Clinical Research Support Team.
Supporting Information: Study Protocol
Time Frame: immediately following publication. no end date.
Access Criteria: Anyone who wishes to access the data. any purpose. Data are available indefinitely.